CLINICAL TRIAL: NCT05182541
Title: Psychological Screening and Nursing of Twin Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Principal Investigator, Caixia Liu, Clinical Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PST in TP
Record Dates: First submitted 2021-06-27; First posted 2022-01-10 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Twin; Complicating Pregnancy; Psychology
Keywords: Twin pregnancy; Psychological screening; nursing
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided self help (Experimental): Introduce the knowledge about twins pregnancy, and reduce the pregnant stress, and relief the anxiety and depressor.
  Interventions: Other: Guided self help; Other: Problem solving therapy
- Face to face PST course (Experimental): Problem cognition and emotional response guidance
  Interventions: Other: Problem solving therapy; Other: Face to face PST course
- Professional psychological intervention (Experimental): Give the pregnancy woman the professional psychological intervention
  Interventions: Other: Professional psychological intervention

INTERVENTIONS:
Other: Guided self help — Introduce the knowledge about twins pregnancy, and reduce the pregnant stress, and relief the anxiety and depressor.
  Arms: Guided self help
Other: Problem solving therapy — Based on the steps of problem-solving therapy, nurses guide mothers with mild psychological problems to solve the existing problems through wechat and telephone, 10-15 min each time for 4 weeks
  Arms: Face to face PST course; Guided self help
Other: Face to face PST course — Face to face interviews with nurses with psychological counselors, combined with auxiliary tools, identify patients' problems, set goals for patients, provide different solutions, and let patients choose appropriate ways according to their preferences. Once a week, 1 hour for the first time and 45 min for the rest for 5 weeks.
  Arms: Face to face PST course
Other: Professional psychological intervention — The mental health physicians and (or) psychological counselors strengthened the intervention and carried out specialized nursing
  Arms: Professional psychological intervention

SUMMARY:
Objectives This research will screen the psychological problems of twin pregnant women step by step and detect early and treat early in order to reduce the incidence of mental diseases and promote the health of mother and baby.

DETAILED DESCRIPTION:
Method Twin pregnant women recruited for the study.The two groups were given routine treatment and nursing measures. The trained group members were given routine psychological care to the control group, while the intervention group was given step-by-step psychological care at the same time.

Evaluate the effect

1. Evaluation methods include process evaluation and result evaluation. Process assessment means that the researchers use the pregnancy stress scale, self rating depression scale and self rating anxiety scale to assess the stress, anxiety and depression of patients at different stages, and make intervention decisions according to the score results; Results evaluation means that if the intervention is effective at a certain stage, the researcher can use it again
2. The evaluation indexes included PPS / SAS / SDS, incidence of preterm birth, premature rupture of membranes and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of intrauterine twin pregnancy.
* The patients whose psychological screening scale score reached the critical value (pregnancy stress scale >50 and/or Self rating depression scale ≥ 40 and/or The self rating Anxiety Scale (SAS) was more than 50.
* The outpatient department of the research hospital was established and antenatal examination was carried out regularly.
* No mental and communication disorders (including depression and other mental diseases).
* Voluntary participation in this study

Exclusion Criteria:

* Pregnancy complicated with severe physical diseases;
* Drop out of this study due to various reasons (including abortion, unwilling to participate in this study)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pregnancy stress scale Self rating Anxiety Scale Depression self rating scale（PPS/SAS/SDS） | pregnancy 6-14 week
  If scores are less than 50, it is defined as normal; If scores are 50-59, it is defined as mild pregnancy stress; If scores are 60-69, it is defined as moderate pressure; If scores are ≥70, it is defined as severe pregnancy stress
Self-rating Anxiety Scale (SAS) | pregnancy 6-14 week
  If scores are less than 50, it is defined as normal; If scores are 50-59, it is defined as mild anxiety; If scores are 60-69, it is defined as moderate anxiety; If scores are ≥70, it is defined as severe anxiety.
Self-rating Depression Scale (SDS) | pregnancy 6-14 week
  If scores are less than 50, it is defined as normal; If scores are 50-59, it is defined as mild depression; If scores are 60-69, it is defined as moderate depression; If scores are ≥70, it is defined as severe depression

SECONDARY OUTCOMES:
Self-rating Anxiety Scale (SAS) | 28-37 weeks; after delivery 1 month
  If scores are less than 50, it is defined as normal; If scores are 50-59, it is defined as mild anxiety; If scores are 60-69, it is defined as moderate anxiety; If scores are ≥70, it is defined as severe anxiety.
Self-rating Depression Scale (SDS) | 28-37 weeks; after delivery 1 month
  If scores are less than 50, it is defined as normal; If scores are 50-59, it is defined as mild depression; If scores are 60-69, it is defined as moderate depression; If scores are ≥70, it is defined as severe depression
Pregnancy stress scale | 28-37 weeks; after delivery 1 month
  If scores are less than 50, it is defined as normal; If scores are50-59, it is defined as mild pregnancy stress; If scores are 60-69, it is defined as moderate pressure; If scores are ≥70, it is defined as severe pregnancy stress
Gestational age and prolongation of gestational age at delivery | 28-37 weeks; after delivery 1 month
  Gestational age at which symptoms of preterm birth occur and gestational age at delivery after treatment
Weight in kilogram of neonate | At birth of neonate
  measured by nurses

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
Research results and conclusions